CLINICAL TRIAL: NCT02627092
Title: An Innovative Approach to Understanding and Controlling Transmission of HAIs
Brief Title: IMPACT STUDY: Investigating Microbial Pathogen Activity of Copper Textiles
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 822418
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Copper linen exposure (Experimental): Subjects will use copper linens during their hospital stay, consisting of copper hospital gowns, copper bed sheets (top and bottom sheets), and copper pillow covers.
  A subset of 50 subjects from this arm will be recruited to provide three types of swabs to calculate the microbial burden on copper linens. Linen swabs, anatomical swabs and environmental swabs will be collected from subjects and subject hospital rooms will be collected to do bacteria counts.
  Interventions: Other: Copper linen exposure
- Non-copper linen exposure (No Intervention): Subjects will not have exposure to copper linens during their hospital stay. They will use the usual hospital linens provided by hospital, not containing copper.
  A subset of 50 subjects from this arm will be recruited to provide three types of swabs to calculate the microbial burden on copper linens. Linen swabs, anatomical swabs and environmental swabs will be collected from subjects and subject hospital rooms will be collected to do bacteria counts.

INTERVENTIONS:
Other: Copper linen exposure — Subjects will use hospital linens (top sheet, bottom sheet, pillow case, gown) made with copper to see if this helps reduce infections during their hospital stay.
  Arms: Copper linen exposure

SUMMARY:
The purpose of this study is to assess the impact of copper linens on hospital acquired infections and drug resistant bacteria.

DETAILED DESCRIPTION:
Healthcare-associated infections (HAIs), particularly those due to multidrug-resistant organisms (MDROs), are of great clinical and public health concern. Although evidence-based prevention strategies have resulted in some success in curtailing HAIs, novel approaches are needed to achieve further reductions. Efforts to curb the emergence of MDROs have been largely unsuccessful. Thus, new strategies to address MDROs are urgently needed. This grant is comprised of two complementary studies that focus on identifying innovative approaches to more effectively prevent HAIs and curtail further emergence of MDROs.

We will conduct a randomized controlled trial (RCT) to assess the efficacy of copper oxide-impregnated textiles in preventing HAIs and MDROs as well as in reducing environmental microbial contamination. We hope to provide critical information to inform the development of novel strategies, and enhance the impact of existing strategies, to successfully address HAIs and MDROs.

For approximately four months the hospital is conducting a research study to learn about the possible impact of copper linens in reducing hospital acquired infections. Some rooms will have copper linens (Group 1) and some rooms will have regular linens (Group 2). The linens will be comprised of the top and bottom sheets, pillowcase cover, and hospital gown.

Patients in both groups will be asked to provide samples during their stay in the ICU. For both study groups, the linens will be sampled twice after they are placed. This will occur on 2 consecutive days. At the same time, study staff will take samples from several areas of the room (the hand rails, overbed table, nurse call button).

Patients will also be asked to allow the research team to obtain swabs of the nose, per-rectal area, armpit and groin. These swabs will be performed on their first day enrolled into the study, then 4 days later, and every week until ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Hospital inpatients
* Admission to intensive care unit
* Hospital Admission at least 48 hours

Exclusion Criteria:

* Hospital admission less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Assessment of intensive care -related hospital-acquired infections or multi-drug resistant organisms | Duration of ICU (must be >48 hours) stay plus 2 additional hospital days
  Number of positive ICU-related MDRO cultures (Methicillin-resistant Staphylococcus aureus or MRSA, Vancomycin-resistant enterococcus or VRE, Carbapenem-resistant Enterobacteriaceae or CRE, Extended-spectrum beta-lactamase or ESBL, Clostridium difficile or C.diff)

CONTACTS AND LOCATIONS:
Overall Officials: Ebbing Lautenbach, MD,MPH,MSCE, Principal Investigator — Univeristy of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No data will be shared.